CLINICAL TRIAL: NCT05806905
Title: Epidemiology, Clinical Features and Diagnosis of Spondylodiscitis at Assiut University Hospital
Brief Title: Spondylodiscitis Cases at Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Osama Ahmed Ibrahiem, Principal investigator, Assiut University
Other Study IDs: ECFDSAUH
Record Dates: First submitted 2023-03-25; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Spondylodiscitis
MeSH Terms: conditions — Discitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The term Spondylodiscitis (SD) involves infection of the vertebra (Spondylitis), infection of the intervertebral disc (Discitis), or both (Spondylodiscitis) Spondylodiscitis is a rare disease accounting for 2.7% of all cases of pyogenic osteomyelitis, with incidence varying from 1 per 100,000/year to 1 per 250,000/year However, there is evidence that the incidence is rising due to longer life expectancy for patients with increasing incidence of chronic debilitating disease including diabetes mellitus, malignancies ,(Human Immunodeficiency Virus (HIV)/ Acquired Immunodeficiency Syndrome (AIDs) , immunosuppressive therapy, increasing numbers of Intravenous drug users , and spinal surgeries.

Pathogens can reach the spine either by: hematogenous spread, direct external inoculation, or spread from contiguous tissues harboring these pathogens. The hematogenous route is the predominant one, allowing seeding of infection from distant sites into the vertebral column.

Since spondylodiscitis has not been studied in a clinical trial at our hospital, and information about this disease has come from retrospective case series and isolated cases. In this study, we present our prospectively collected patient clinical and epidemiological data in order to provide a proper management

ELIGIBILITY:
Inclusion Criteria:

* All patients who come into Assiut University Hospital and outpatient clinic with clinical symptoms suggestive of spondylodiscitis in all age groups including patients with known medical conditions and patients who underwent previous spine surgeries (post operative spondylodiscitis)

Exclusion Criteria:

* No patients will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who come into Assiut University Hospital and outpatient clinic with clinical symptoms and radiological findings suggestive of spondylodiscitis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
measuring the inflammatory markers in patient with spondylodiscitis (Ex. C reactive protein (CRP) in mg/dl) | collect data for 1 year and follow up for 1 year
  collect all patients with spondylodiscitis who come to Assiut University Hospital, measure the inflammatory markers and follow up them after medical or surgical treatment
Describing of pain severity according to Pain severity scale and follow up after treatment | collect data for 1 year and follow up for 1 year
  collect all patients with spondylodiscitis who come to Assiut University Hospital, measure the pain severity and follow up pain improvement after medical or surgical treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Kamal AM, El-Sharkawi MM, El-Sabrout M, Hassan MG. Spondylodiscitis: experience of surgical management of complicated cases after failed antibiotic treatment. SICOT J. 2020;6:5. doi: 10.1051/sicotj/2020002. Epub 2020 Feb 14. PMID 32057290
- [Background] D'Agostino C, Scorzolini L, Massetti AP, Carnevalini M, d'Ettorre G, Venditti M, Vullo V, Orsi GB. A seven-year prospective study on spondylodiscitis: epidemiological and microbiological features. Infection. 2010 Apr;38(2):102-7. doi: 10.1007/s15010-009-9340-8. Epub 2010 Feb 27. PMID 20191397
- [Background] Kaya S, Kaya S, Kavak S, Comoglu S. A disease that is difficult to diagnose and treat: evaluation of 343 spondylodiscitis cases. J Int Med Res. 2021 Nov;49(11):3000605211060197. doi: 10.1177/03000605211060197. PMID 34851766
- [Background] Issa K, Diebo BG, Faloon M, Naziri Q, Pourtaheri S, Paulino CB, Emami A. The Epidemiology of Vertebral Osteomyelitis in the United States From 1998 to 2013. Clin Spine Surg. 2018 Mar;31(2):E102-E108. doi: 10.1097/BSD.0000000000000597. PMID 29135608
- [Background] Gerometta A, Bittan F, Rodriguez Olaverri JC. Postoperative spondilodiscitis. Int Orthop. 2012 Feb;36(2):433-8. doi: 10.1007/s00264-011-1442-0. Epub 2012 Feb 4. PMID 22307558
- [Background] Sur A, Tsang K, Brown M, Tzerakis N. Management of adult spontaneous spondylodiscitis and its rising incidence. Ann R Coll Surg Engl. 2015 Sep;97(6):451-5. doi: 10.1308/rcsann.2015.0009. Epub 2015 Aug 14. PMID 26274746
- [Background] Turgut M. Complete recovery of acute paraplegia due to pyogenic thoracic spondylodiscitis with an epidural abscess. Acta Neurochir (Wien). 2008 Apr;150(4):381-6. doi: 10.1007/s00701-007-1485-6. Epub 2008 Jan 8. PMID 18176773